CLINICAL TRIAL: NCT05519943
Title: Effectiveness of Group CBT on Internalizing and Externalizing Symptoms in Children With Mixed Psychiatric Disorders
Brief Title: Effectiveness of Group CBT in Children With Mixed Psychiatric Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Sarianna Barron-Linnankoski, Principal Investigator, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/211/2016
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Child Behavior Problem
Keywords: children; group cognitive behavioral therapy; cognitive behavioral therapy; internalizing symptoms; externalizing symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group cognitive behavioral therapy intervention (Experimental)
  Interventions: Behavioral: The Friends program
- Treatment as usual (TAU) (Experimental)
  Interventions: Behavioral: TAU condition

INTERVENTIONS:
Behavioral: The Friends program — A GCBT intervention comprising ten weekly 60-minute sessions followed by two booster sessions
  Arms: group cognitive behavioral therapy intervention
Behavioral: TAU condition — A TAU waitlist condition during which participants received routine care services tailored to each child individually.
  Arms: Treatment as usual (TAU)

SUMMARY:
This study aims to examine the immediate and longer-term effectiveness of a group cognitive behavioral therapy intervention (GCBT) in reducing internalizing and externalizing symptoms in children treated for mixed psychiatric disorders in naturalistic clinical settings. Further, the effectiveness of GCBT is compared to a treatment-as-usual condition (TAU). Within this study, it is hypothesized that children with mixed psychiatric disorders will exhibit improvements in parent-rated internalizing problem behavior and parent- and teacher-rated externalizing problem behavior following GCBT.

ELIGIBILITY:
Inclusion Criteria:

* Helsinki University Hospital child psychiatric outpatient clinic patients with symptoms of anxiety or depression, deficiencies in emotional and behavioral skills impairing functioning, and sufficient social and cognitive skills to participate in group work.

Exclusion Criteria:

* Helsinki University Hospital child psychiatric outpatient clinic patients with excessive physical aggression, excessive physical restlessness to enable skill training, or whose severity of psychiatric symptoms required individual psychotherapy (e.g., acute suicidality or psychosis).

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in parent- and teacher rated internalizing and externalizing symptoms | From referral to GCBT to 6-month follow-up
  The Child Behavior Check List (CBCL) and the Teacher´s Report Form (TRF)

IPD SHARING:
Plan to Share IPD: No